CLINICAL TRIAL: NCT02551978
Title: Kids Obesity Prevention Program - Study (KOP). A Serious Game to Address Barriers to Prevention and Treatment of Obesity in Primary School Children
Brief Title: Kids Obesity Prevention Program - Study (KOP)
Acronym: KOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Science Campus Tuebingen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KOP_1
Record Dates: First submitted 2015-09-11; First posted 2015-09-16 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-09

CONDITIONS: Obesity; Child
Keywords: obesity; child; primary prevention; serious game; nutrition; physical activity; psychosocial; stress; knowledge; diet
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Children in a primary school, aged between 9 and 12 years, play the serious game (two sessions, duration of each session 35 minutes, within two weeks). The game equips the children with knowledge about the core areas nutrition, physical activity, and psychosocial factors.
  Interventions: Other: The serious game KOP
- Control (No Intervention): Children in the same primary school, aged between 9 and 12 years do receive basic information during the study phase.

INTERVENTIONS:
Other: The serious game KOP — The serious game transfers knowledge about nutrition (food pyramid, energy density of foods, which foods contribute to satiety and which not, energy in liquids, self-reflexive diagnostic tool to analyze daily food intake), physical activity (a motion-control to navigate through the game is partly used, relationship between energy expenditure and energy intake) and psychological aspects (relaxation-exercises, what is stress, stress-coping strategies).
  Arms: Intervention

SUMMARY:
Obesity and its associated comorbidities are becoming a key and rapidly growing public health problem. The cause of obesity is an imbalance between energy intake and energy expenditure in favor of the former. Childhood and adolescence are seen as critical time for its development. It is therefore crucial to provide both prevention and treatment actions already during childhood. The prevention and treatment weight-management programs in children focus on improving diet, eating behaviours, psychosocial aspects and increasing physical activity. One important basic requirement for any weight-management program is, that both children and their families are motivated and ready for change. Video games, including exergames, serious games or combined approaches offer additional chances in the treatment and prevention of obesity by approaching children in their environment and motivating them to deal with life-style topics.

The investigators developed a motion-controlled serious game for children aged between 9 and 12 years, addressing all the three core areas nutrition, physical activity, and psychosocial factors. In addition to the motion control, a tablet is used for knowledge-based and cognitive tasks. In comparison to other studies the nutrition part not only deals with the food pyramid but also with the energy density of foods and liquids and offers a self-reflexive diagnostic tool to analyse daily food intake. Moreover, psychological aspects, especially stress and stress-coping strategies are addressed e.g. by relaxation-exercises. The game consists of two sessions, having each a duration of about 35 minutes.

The aim of this study is to evaluate the program in a cluster-randomized controlled trial in a primary school setting in children aged 9 to 12 years. Therefore, six 4th grade classes of the same school will be randomly allocated to an intervention and a control group. The intervention group will play the game within two weeks, whereas the control group will receive basic information. At baseline, two weeks after baseline and at four weeks follow-up, measurements will be performed. The primary outcome of the study is the gain of knowledge (nutrition, psychosocial aspects) measured by a self-constructed questionnaires tailored specifically for the serious game. Secondary outcomes are the acceptance of the game, changes of nutrition behaviour, physical activity and intentions of the children to follow a healthy lifestyle, measured by mostly validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* all children which belong to the 4th graders of a primary school

Exclusion Criteria:

* children with massive linguistic difficulties will be excluded (after study participation; due to ethical reasons we can not do this ahead)

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Knowledge of the children about nutrition and psychosocial aspects by a self-developed questionnaire specific for the serious game | Change between baseline and two weeks after the baseline measurement

SECONDARY OUTCOMES:
Nutrition Score (Ernährungsmusterindex) by Kleiser et al., 2007 used in the KIGGS cohort (Studie zur Gesundheit von Kindern und Jugendlichen in Deutschland) | Change between baseline and four weeks follow-up (on average 6 weeks after baseline measurement))
  Parents and children are independently asked to report the food frequencies for key foods in order to calculate the Ernährungsmuster index
Food frequency of specific foods which are addressed in the serious game | Change between baseline and four weeks follow-up (on average 6 weeks after baseline measurement))
  Parents and children are independently asked to report the food frequencies of specific foods
Physical activity using a validated questionnaire filled in by the children and also the parents | change between baseline and four weeks follow-up (on average 6 weeks after baseline measurement))
  Parents and children are independently asked to fill in the questionnaire
Intentions of children to stick to a healthy lifestyle by using a tailored questionnaire specific for the contents of the serious game | Change between baseline, and two weeks after baseline measurement, and four weeks follow-up
Acceptance of the serious game by the children using a self-developed questionnaire specific for the serious game | At baseline and directly after the end of the second session of the game (on average two weeks after baseline measurement)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Zipfel, Prof. Dr., Principal Investigator — University Hospital Tuebingen, Germany

REFERENCES:
- [Derived] Mack I, Reiband N, Etges C, Eichhorn S, Schaeffeler N, Zurstiege G, Gawrilow C, Weimer K, Peeraully R, Teufel M, Blumenstock G, Giel KE, Junne F, Zipfel S. The Kids Obesity Prevention Program: Cluster Randomized Controlled Trial to Evaluate a Serious Game for the Prevention and Treatment of Childhood Obesity. J Med Internet Res. 2020 Apr 24;22(4):e15725. doi: 10.2196/15725. PMID 32329742
- See also: Related Info — http://www.wissenschaftscampus-tuebingen.de